CLINICAL TRIAL: NCT03400020
Title: Efficacy of Vitamin C Administration for the Prevention of Postpolypectomy Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilam University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Assistant Professor, Ilam University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13961019; NCT03374410 (obsolete NCT alias)
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Postpolypectomy Bleeding
MeSH Terms: interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascorbic acid (Experimental): Ascorbic acid 1000 mg in normal saline IV 2 hours before the operation and thereafter 500 mg in normal saline IV daily for three days.
  Interventions: Other: Ascorbic acid
- Normal saline (Placebo Comparator): Normal saline IV infusion 2 hours before the operation and for three days after operation.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Ascorbic acid — Ascorbic acid 500 Mg in normal saline IV two hours before the operation and thereafter 500 mg in normal saline IV daily for three days.
  Other Names: Vitamin C
  Arms: Ascorbic acid
Other: Normal Saline — Normal saline IV two hours before the operation and thereafter for three days.
  Arms: Normal saline

SUMMARY:
Postpolypectomy bleeding is the most common major complication following a colonoscopic polypectomy procedure. The incidence rate ranging from 0.3 to 6.1%. Several preventive methods such as detachable snare and adrenaline injection have been proposed in the management of postpolypectomy bleeding in large colonic polyps. It has been demonstrated that administration of ascorbic acid (vitamin C) in abdominal surgeries could reduce the blood loss during the procedure, operation time and days of hospitalization. So the investigators designed a prospective, randomized study to compares the efficacy of vitamin C administration with application of prophylactic clip and detachable snare in the prevention of postpolypectomy bleeding in large polyps.

DETAILED DESCRIPTION:
In this prospective, randomized clinical trial, patients diagnosed with colon polyps with a diameter > 10 mm will randomized to receive either a 500 mg vitamin C in normal saline injection or a normal saline injection 2 hours before polypectomy. This administration will continued for 3 days after polypectomoy. Postpolypectomy bleeding is defined either as (1) early: occurring either during an endoscopic procedure or immediately after as hematochezia within 24 h or (2) delayed: any bleeding event that occurring between day 2 and day 30 following the polypectomy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal polyps larger than 10 mm.

Exclusion Criteria:

bleeding tendency poor preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Early postpolypectomy bleeding | up to 24 hours
  bleeding occurring either during an endoscopic procedure or immediately after as hematochezia within 24 hours following the polypectomy procedure.
Late postpolypectomy bleeding | between day 2 and day 30
  bleeding occurring between day 2 and day 30 following the polypectomy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shaahin Shahbazi, MD, Study Chair — Ilam University of Medical Sciences
Locations (1):
- Mostafa Khomaini Hospital, Īlām, Iran

IPD SHARING:
Plan to Share IPD: No